CLINICAL TRIAL: NCT05434546
Title: A Randomized, Open-label, Multicenter, Phase 2 Clinical Trial to Explore the Safety and Efficacy of Sepranolone in Pediatric and Adult Patients With Tourette Syndrome
Brief Title: A Study to Explore the Effect of Sepranolone in Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asarina Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APH205
Record Dates: First submitted 2022-03-12; First posted 2022-06-28 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Tourette Syndrome; Tourette Syndrome in Adolescence
Keywords: Tourette Syndrome in Adults
MeSH Terms: conditions — Tourette Syndrome | interventions — Pregnanolone

STUDY DESIGN:
Intervention Model Description: Interventional, open-label, multicenter, randomized, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sepranolone (Experimental): Sepranolone 10 mg sc twice weekly for 12 weeks alongside the patient's standard of care Tourette treatment.
  Interventions: Drug: Sepranolone
- No Intervention (No Intervention): Continuation of the patient's standard of care Tourette treatment for 12 weeks.

INTERVENTIONS:
Drug: Sepranolone — Treatment with 10 mg Sepranolone s.c. twice weekly for 12 weeks alongside patient's standard of care Tourette treatment.
  Other Names: Isoallopregnanolone
  Arms: Sepranolone

SUMMARY:
The study was an open-label, randomized, multicenter, parallel, Phase 2a study in adolescents and adult patients with Tourette syndrome that aimed to explore the efficacy of Sepranolone as a treatment for Tourette syndrome, by reducing the severity and frequency of tics. The total study duration from the Screening Visit to the final follow-up visit was approximately 26 weeks and included the following periods:

* A baseline period of 4 weeks between the screening visit (Visit 1) and randomization (4 weeks of baseline period were not needed in well-known adult subjects with stable Tourette syndrome history over the past at least 4 weeks). A school holiday/annual leave period of 2-6 weeks where no study-related activities were done.
* A randomized treatment period of 12 weeks
* A safety follow-up period of 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Tic severity score ≥ 20 Yale Global Tic Severity Scale (YGTSS) Total Score at baseline
* The patient may have Obsessive-Compulsive Disease (OCD) as a comorbidity

Exclusion Criteria:

* Patient has participated in a clinical study over the past 30 days
* Evidence or history of neurological disease that may interfere with the study
* Malignant disease
* Unstable or clinical significant medical condition that could pose a risk
* HIV/ongoing hepatitis
* Clinical significant findings in vital signs
* History of anaphylactic reactions

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of Sepranolone to reduce tic severity in patients with Tourette syndrome at 12 weeks, as measured by change in baseline in the The Yale Global Tic Severity Scale (YGTSS) Total Score. | Change from baseline at week 4, 8 and 12.
  The Yale Global Tic Severity Scale (YGTSS) is a validated scale for assessing the severity of motor and vocal tics in both children and adults with Tourette syndrome. Tics are scored based on a semi-structured interview, including scoring of the number, frequency, intensity, complexity, and interference of tics. The primary endpoint is the total tic score assessment. The score ranges from 0-50, where a higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Safety and tolerability of Sepranolone in adolescent and adult patients with Tourette syndrome | From randomization (day 1) until the end of study visit (week 16).
  Collection of adverse events (AEs) including spontaneous reporting, number of subjects with clinically significant changes in clinical safety laboratory blood and urine test values, vital signs, weight, and injection related events.
To evaluate the efficacy of Sepranolone to reduce tic related impairment in patients with Tourette syndrome at 12 weeks, as measured by change in baseline in the Yale Global Tic Severity Scale (YGTSS) Impairment Score. | Change from baseline at week 4, 8 and 12.
  The Yale Global Tic Severity Scale (YGTSS) is a validated scale for assessing the severity of motor and vocal tics in both children and adults with Tourette syndrome. Tics are scored based on a semi-structured interview, including scoring of the number, frequency, intensity, complexity, and interference of tics. The secondary endpoint is the impairment score assessment. The score ranges from 0-50, where a higher score indicates a worse outcome.
To evaluate the efficacy of Sepranolone to reduce the urge to tic in patients with Tourette syndrome at 12 weeks, as measured by change in baseline in the Premonitory Urge for Tics Scale (PUTS) scale. | Change from baseline at week 4, 8 and 12.
  The Premonitory Urge for Tics Scale (PUTS) scale is an assessment aiming to quantify the premonitory urge to tic. The scale is reliable and valid instrument for children from above the age of 10 and for adults. This scale is used as a self-report assessment instrument, where the Investigator asks 10 questions, out of which the score for the first 9 questions add up to the total score (i.e., the 9-Item Total). The respondent has 4 alternatives, "not at all true", "a little true", "pretty much true" and "very much true," represented by a score or 1-4, respectively. The total score ranges from 9-36, where a higher score indicates a worse outcome.
To evaluate the effect of Sepranolone on activities of daily living in patients with Tourette syndrome at 12 weeks, as measured by change in baseline in the GTS-QoL ADL subscale. | Change from baseline at week 4, 8 and 12.
  The Gilles de la Tourette Syndrome - Quality of Life (GTS-QoL) physical/activities of daily living (ADL) subscale assesses the impact of the symptoms of Tourette syndrome on the subject's quality of life. The instrument consists of 27 questions, asked by an interviewer, where subjects score the extent of impact on a 5-point verbal scale ranging from "no problems" to "extreme problems." The score ranges from 27-135, where a higher score indicates a worse outcome.
To evaluate the effect on Global impression by Sepranolone in patients with Tourette syndrome at 12 weeks, as measured by the Tourette Syndrome-Clinical Global Impression (TS-CGI). | TS-CGI score at week 4, 8 and 12.
  The Tourette Syndrome-Clinical Global Impression (TS-CGI) is a clinician rating of the change in severity of the symptoms of Tourette syndrome. The scale is a 7-step Likert scale, where the following alternatives are represented by a score of 1-7, respectively: "very much worsened," "much worsened," "minimally worsened," "no change," "minimally improved," "much improved," or "very much improved." The score ranges from 1-7, where a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Debes, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (2):
- Denmark (2):
  - Herlev Hospital, Copenhagen, Herlev
  - Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No